CLINICAL TRIAL: NCT00813332
Title: A Double Blind , Randomized, Multicenter Study of Second Line Treatment of Endostar（rh Recombined Endostatin）With Single Docetaxel In NSCLC Patients
Brief Title: Second-line Therapy Study of Combined Chemotherapy and Endostar to Patients With Non-Small Cell Lung Cancer(NSCLC)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Simcere Pharmaceutical Co., Ltd (Other)
Responsible Party: Kai LI/Professor, Cancer Hospital of Tianjin Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: simcere002; simcere0802
Record Dates: First submitted 2008-12-19; First posted 2008-12-23 (Estimated); Last update posted 2010-01-25 (Estimated); Status verified 2009-12

CONDITIONS: Advanced NSCLC; Recurrent NSCLC
Keywords: Endostar; NSCLC; Docetaxel; Combined therapy; second-line chemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel; Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Endostar combined with Docetaxel for Advanced NSCLC: All eligible patients will receive Endostar in combination with Docetaxel chemotherapy for 2 cycles (21 days for each cycle) and cases of good response(CR+PR+SD) will continue treatment for 2 cycles. Endostar treatment will continue after completion of first 4 cycles until disease progression.
  Interventions: Drug: Endostar(rh recombinant endostatin) plus Docetaxel
- 2 (Placebo Comparator): Docetaxel combined with placebo for Advanced NSCLC: All eligible patients will receive placebo in combination with Docetaxel chemotherapy for 2 cycles (21 days for each cycle) and cases of good response(CR+PR+SD) will continue treatment for 2 cycles. Placebo will continue after completion of first 4 cycles until disease progression.
  Interventions: Drug: Placebo plus Docetaxel

INTERVENTIONS:
Drug: Endostar(rh recombinant endostatin) plus Docetaxel — 7.5mg/m2, IV( in the vein) on day1-14 of each 21-28 day cycle. Number of cycles: until progression or unacceptable toxicity develops.
  Other Names: Experimental group
  Arms: 1
Drug: Placebo plus Docetaxel — Placebo plus Docetaxel
  Other Names: control group
  Arms: 2

SUMMARY:
The purpose of this study is to compare the efficacy and safety of Endostar (Recombinant Human Endostatin) combined with Docetaxel and single Docetaxel through multi-center, double-blinding, randomized controlled, phase Ⅳ clinical trial for NSCLC cases who have obvious progressive disease or intolerant adverse effects in first-line chemotherapy.

DETAILED DESCRIPTION:
The combinative therapy of Endostar, Vinorelbine and cisplatin has been shown to increase response rate and survival in patients (pts) with advanced NSCLC and is sFDA-approved for this indication. However, there are limited data on the safety and efficacy of Endostar in combination with other widely used chemotherapy doublets for NSCLC. Clinical data proved that Endostar was a wild spectrum and safe antiangiogenesis factor which could suppress almost 65 kinds of tumor mass in animal models and affect about 12 percent human genome. In this clinical trial, there will be 160 patients enrollment, giving Docetaxel (75mg/m2,iv, d1, every 3 weeks) plus Endostar(7.5mg/m2/day, iv, d1-d14, every 3 weeks) or Docetaxel with placebo. We'll evaluate the efficacy and safety of the Docetaxel plus Endostar treatment to NSCLC and hope to provide a promising regimen to advanced lung cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old, males or females;
2. Patients with NSCLC confirmed by histopathology or cytology who need second-line chemotherapy, including progressive disease cases during or in 3 months posterior to end of first-line chemotherapy( at least 4 cycles done) and cases with intolerant adverse effects in first-line chemotherapy( at least 4 cycles done); neo-adjuvant chemotherapy and targeted therapy(EFGR-TKIs) not to be served as first-line chemotherapy; 3 months of clearance needed for neo-adjuvant chemotherapy and 1 month for targeted and first-line chemotherapy;
3. Local advanced and metastatic cases with tumor foci that can be evaluated by CT, MRI or PET-CT; at least one diameter ≥ 1 cm (including metastatic lymph nodes) confirmed by CT scan or ≥ 1 cm by spin CT or PET-CT );
4. No contraindication for chemotherapy, with normal peripheral hemogram, renal and hepatic function: Peripheral hemogram: WBC≥4.0×109/L，PLT≥80×109/L，Hgb≥90g/L； Renal function: serum BUN and creatinine ≤1.0×UNL; Hepatic function: transaminase≤1.5×UNL, BIL≤×UNL;
5. Karnofsky performance scale≥60 or ECOG performance scale≤ 2; expected survival time≥3 months;
6. No allergic history to biological agents and taxane agents;
7. Patients are voluntary to participate and sign the informed contents.

Exclusion Criteria:

1. Pregnant or breast-feeding females; or females who have reproductive ability but do not take contraception method;
2. With severe acute infection uncontrolled; purulent or chronic infection with wounds difficult to recover;
3. With history of severe heart diseases, including congestive heart failure, uncontrolled arrhythmia with high risk, unstable angina pectoris, myocardial infarction, severe cardiac valvular diseases and refractory hypertension;
4. Patients with uncontrolled neurological, mental disease or psychosis, patients with poor compliance that cannot coordinate the therapy or describe the treatment response;
5. Uncontrolled brain metastasis patients with obvious manifestations of intracranial hypertension or neurological and mental disorders;
6. Uncontrolled diabetes and contraindication to corticoid agents;
7. Obvious hemorrhage tendency;
8. Allergic to any drug in the trial;
9. Patients with a second tumor;
10. Patients participating in other clinical trials;
11. Patients treated by Endostar or Docetaxel (excluding neo-chemotherapy) included combination chemotherapy previously;
12. Foci to be evaluated for response in trial treated by radiation in 6 months.
13. Other conditions that are regarded for exclusion by the trialists.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2008-10; Primary Completion 2009-10 (Estimated); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival time,survival rate for 1 year | two years (2010.10)

SECONDARY OUTCOMES:
Tumor response rate, disease controlled rate and adverse effects. | 1 year (2009.10)

CONTACTS AND LOCATIONS:
Overall Officials: Kai LI, professor, Principal Investigator — Cancer Hospital of Tianjin Medical University
Locations (1):
- Cancer Hospital of Tianjin Medical University, Tianjin, China